CLINICAL TRIAL: NCT01968616
Title: Predictive Factors of 2-year Visual Outcome in Retinal Vein Occlusion Following Intravitreal Ranibizumab Treatment
Brief Title: Ranibizumab Treatment for Retinal Vein Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Nagahisa Yoshimura, Department of Ophthalmology & Visual Sciences, Kyoto University, Graduate School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-RV-R
Record Dates: First submitted 2013-10-20; First posted 2013-10-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Macular Edema Due to BRVO/CRVO
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Lucentis 0.5mg (Other): One arm
  Interventions: Drug: Ranibizumab, 0.5mg, Intravitreal

INTERVENTIONS:
Drug: Ranibizumab, 0.5mg, Intravitreal

SUMMARY:
In retinal vein occlusion, predictive factors for visual outcome after ranibizumab treatment have not been evaluated comprehensively. Therefore, we have planned to analyze predictors for visual outcome from a viewpoint of electrophysiology and biomarkers besides morphological features by SD-OCT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Male or female of aged 18 years or older
* Macula edema secondary to BRVO/CRVO
* Decrease of VA due to macular edema

Exclusion Criteria:

* Prior episode of RVO
* Previous treatment with anti-VEGF drugs or corticosteroid or grid laser photocoagulation (study eye)
* Ocular disorders in the study eye that may confound interpretation of study results
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for RVO
* The pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Mean foveal thickness measured by SD-OCT | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Kyoto University Hospital, Kyoto, Kyoto, Japan